CLINICAL TRIAL: NCT01794585
Title: Home-Based Virtual Reality (VR) Treatment for Chronic Balance Problems in Adults With Traumatic Brain Injury
Brief Title: Virtual Reality (VR) Treatment for Balance Problems in Traumatic Brain Injury (TBI)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Craig Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H133A120032-2
Record Dates: First submitted 2012-11-12; First posted 2013-02-20 (Estimated); Last update posted 2018-02-06 (Actual); Status verified 2018-02

CONDITIONS: Traumatic Brain Injury
Keywords: traumatic brain injury; balance deficits; virtual reality; home-based therapy
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Virtual Reality Based Exercise (Experimental)
  Interventions: Behavioral: Virtual Reality Based Exercise
- Standard Exercise (Active Comparator)
  Interventions: Behavioral: Standard Exercise

INTERVENTIONS:
Behavioral: Virtual Reality Based Exercise — A structured, individually tailored, protocol driven, reproducible therapeutic intervention. The study intervention will consist of individually prescribed selections from three off-the-shelf VR games that target the type and severity of balance deficits elicited during the completion of a baseline assessment. Participants randomized to receive this intervention will be assigned a home balance program that utilizes an Xbox Kinect system to provide balance activities.
  Arms: Virtual Reality Based Exercise
Behavioral: Standard Exercise — An individualized home balance exercise program that also targets identified balance system-specific deficits, however, utilizes no VR components.
  Arms: Standard Exercise

SUMMARY:
The purpose of this study is to evaluate the effectivenes of a home-based physical therapy program designed to improve balance following traumatic brain injury by incorporating the use of a virtual reality system.

ELIGIBILITY:
Inclusion Criteria:

* Has sustained a documented TBI that required an inpatient rehabilitation program;
* is at least one year post TBI;
* is at least 18 and no more than 64 years of age at the time of enrollment;
* is English or Spanish speaking
* is at least three months beyond completion of formal PT, including acute inpatient rehabilitation, outpatient and home-based therapy;
* provides written medical clearance for participation in an in-home balance exercise program;
* ambulates independently within the home (with assistive devices and/or orthotics as needed);
* has active range of motion of bilateral upper extremities of at least 90 degrees of abduction to allow for control of the VR system;
* completes a 15 minute trial using a VR system in the absence of a negative physical or behavioral reaction;
* self-reports ongoing balance deficits and demonstrate such deficits by scoring at or below one standard deviation above the mean (75 or below) on the CB&M; and
* provides informed consent, or has a guardian available to provide consent.

Exclusion Criteria:

* has a history of another medical illness or neurological disorder which may affect balance;
* has experienced a seizure within the last year;
* has a history of psychiatric disorder requiring hospitalization;
* is currently participating in another RCT;
* is currently using VR technology to address specific balance goals;
* is unable to travel to Craig for assessments throughout the study period;
* is unable to communicate effectively to complete standardized assessments;
* has cognitive impairment that precludes completion of baseline testing;
* is unavailable to participate in 12 continuous weeks of therapy;
* has no access to television able to connect to VR-gaming system; and
* reports inadequate space required for VR-gaming system sensors.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2013-04; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Change from Baseline on Community Balance and Mobility (CB&M) | Baseline, 6-weeks, 12 weeks, 24weeks
  Specifically developed to assess balance function for individuals with TBI. Includes 13 balance based activites such as single leg standing, tandem walking, hopping, running, descending stairs.

SECONDARY OUTCOMES:
Change from Baseline on Balance Evaluation Systems Test (BESTest) | Baseline, 6weeks, 12weeks, 24weeks
  Used to evaluate balance system function. Movement characteristics and timed criteria are used to rate 36 items on a scale of 0 (maximum limitation) to 3 (within normal limits).
Change from Baseline on Activity-specific, Behavior Confidence Scale (ABC) | Baseline, 6weeks, 12weeks, 24weeks
  Used to assess fear of falling, the ABC scale includes 16 items that describe everyday community activities and which are scored on a scale of 0 (no confidence) to 100 (complete confidence).
Change from Baseline on Participation Assessment with Recombined Tools-Objective (PART-O) | Baseline, 6 weeks, 12weeks, 24weeks
  This 17-item assessment of community participation will be used to measure overall societal participation.

CONTACTS AND LOCATIONS:
Locations (1):
- Craig Hospital, Englewood, Colorado, United States

REFERENCES:
- [Derived] Tefertiller C, Hays K, Natale A, O'Dell D, Ketchum J, Sevigny M, Eagye CB, Philippus A, Harrison-Felix C. Results From a Randomized Controlled Trial to Address Balance Deficits After Traumatic Brain Injury. Arch Phys Med Rehabil. 2019 Aug;100(8):1409-1416. doi: 10.1016/j.apmr.2019.03.015. Epub 2019 Apr 19. PMID 31009598